CLINICAL TRIAL: NCT03353818
Title: Golf and Diabetes Can an Introctionary Course to Golf and a Free 1-year Membership in a Golf Club Increase Physichal Activity?
Brief Title: Golf and Diabetes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexander Christensen (Other)
Collaborators: Research Unit for General Practice, Aarhus University (Other)
Responsible Party: Sponsor-Investigator, Alexander Christensen, MD, ph.d.-student, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-17001697
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — GOLF protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Golf (Active Comparator): In three different golf clubs patients will be introduced how to play golf. They will be taught techniques and recieve basic golf equipment. A total of 1 year membership free membership in the golf clubs will be given.
  Interventions: Behavioral: Golf
- Placebo (Placebo Comparator): No intervention given. No restrictions on physical activity.
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Golf — A free golf course and free membership for one year in a golf club will be given to participants.
  Arms: Golf
Behavioral: No intervention — Patients acting as controls will not be restricted in any ways.
  Arms: Placebo

SUMMARY:
This a randomised, single-blinded, controlled study that investigate if a free golf training programme will increase the physical activity of type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2-diabetes
* Physical activity less than 8000 steps per day
* Age > 18 years

Exclusion Criteria:

* Pregnancy
* Conditions that makes patients unfit for participation in golf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Evaluated at baseline and after 6 and 12 months
  Change in physical activity level from baseline to end of study evaluated by 7-days wear of accelerometers.

SECONDARY OUTCOMES:
Quality of life | Evaluated at baseline and after 6 and 12 months
  Use of validated questionaries to evaluate impact of quality of life
Hand muscle strength | Evaluated at baseline and after 6 and 12 months
  Change in hand muscle strength
Diabetic control | Evaluated at baseline and after 6 and 12 months
  Changes in diabetes related biochemistry and cardiovascular risk factors
Adherence | Evaluated at baseline and after 6 and 12 months
  Adherence evaluated with diarries
Estimated VO2max | Evaluated at baseline and after 6 and 12 months
  Two point bicycle test, where an estimated VO2 max can be calculated

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Public Health, Research Unit and Section of General Practice, University of Aarhus, ,, Aarhus
  - Center for Diabetes Research, Gentofte Hospital, Hellerup

IPD SHARING:
Plan to Share IPD: No